CLINICAL TRIAL: NCT02360878
Title: The Endocrine Impact of the Duodenal-jejunal Bypass Sleeve on Type 2 Diabetes - Potential Role of the Incretin Hormones
Status: Completed | Type: Observational
Sponsor: Filip Krag Knop (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Filip Krag Knop, MD, Ph.D., University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Other Study IDs: DJBS meal test
Record Dates: First submitted 2015-01-28; First posted 2015-02-11 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: DJBS; Duodenal-jejunal bypass sleeve; Duodenal-jejunal bypass liner; Endobarrier; Obesity; Type 2 diabetes; Incretin hormones; Postprandial glucose metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood feces
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-diabetic subjects: Obese (BMI > 30 kg/m2) with normal glucose tolerance implanted with the EndoBarrier Gastrointestinal liner
  Interventions: Device: EndoBarrier Gastrointestinal Liner
- T2DM subjects: Obese (BMI > 30 kg/m2) with type 2 diabetes implanted with the EndoBarrier Gastrointestinal liner
  Interventions: Device: EndoBarrier Gastrointestinal Liner

INTERVENTIONS:
Device: EndoBarrier Gastrointestinal Liner — Implantation with the EndoBarrier
  Other Names: DJBS

SUMMARY:
We want to evaluate the impact of the EndoBarrier Gastrointestinal Liner (DJBS) on glucose metabolism as well as gut and pancreatic hormone secretion.

DETAILED DESCRIPTION:
Duodenal-jejunal bypass sleeve (DJBS) is being developed for the treatment of obesity, and initial clinical outcomes suggest that this minimally invasive endoscopic technique potentially has beneficial effects on type 2 diabetes also. However, the mechanisms behind the antidiabetic effects of the procedure remain unknown. We want to elucidate how the DJBS might change postprandial secretion of gut and pancreatic hormones.

ELIGIBILITY:
Inclusion Criteria (obese subjects with type 2 diabetes):

* treatment with DJBS
* written informed consent
* antidiabetic monotherapy/or diet
* > 18 years old
* not anemic

Exclusion Criteria (obese subjects with type 2 diabetes):

* antidiabetic treatment with insulin, GLP-1-agonists, DPP4-inhibitors or more than one orally administered antidiabetic drug.
* anemia

Inclusion Criteria (obese subjects without type 2 diabetes):

* Treatment with DJBS
* written informed consent
* not anemic
* HbA1c < 6,0% or HbA1c < 6,5% and normal glucose tolerance test and normal fasting plasma glucose (< 6,0 mM)

Exclusion Criteria (obese subjects without type 2 diabetes):

* HbA1c > 6,5 % and/or a non-normal glucose tolerance test and/or fasting plasma glucose > 6,0 mM

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese subjects with or without type 2 diabetes treated with the DJBS will be suitable for participating in the trial
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-02; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in postprandial glucagon-like peptide-1 (GLP-1) secretion from baseline 1 week after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucagon-like peptide-1 (GLP-1) secretion from baseline 26 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucagon-like peptide-1 (GLP-1) secretion from baseline 52 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucagon-like peptide-1 (GLP-1) secretion from baseline 3 weeks after explantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes

SECONDARY OUTCOMES:
Change in basal metabolic rate from baseline 1 week after implantation | 0, 50, 210 minutes
Change in basal metabolic rate from baseline 26 weeks after implantation | 0, 50, 210 minutes
Change in basal metabolic rate from baseline 52 weeks after implantation | 0, 50, 210 minutes
Change in basal metabolic rate from baseline 3 weeks after explantation | 0, 50, 210 minutes
Change in gastric emptying from baseline 1 week after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in gastric emptying from baseline 26 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in gastric emptying from baseline 52 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in gastric emptying from baseline 3 weeks after explantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in gallbladder emptying from baseline 1 week after implantation | 0, 20, 40, 60, 90, 120, 150, 180
Change in gallbladder emptying from baseline 26 weeks after implantation | 0, 20, 40, 60, 90, 120, 150, 180
Change in gallbladder emptying from baseline 52 weeks after implantation | 0, 20, 40, 60, 90, 120, 150, 180
Change in gallbladder emptying from baseline 3 weeks after explantation | 0, 20, 40, 60, 90, 120, 150, 180
Change in satiety scores as measured by Visual Analogue Scales 1 week after implantation | 0, 30, 60, 90, 120, 180, 240
Change in satiety scores as measured by Visual Analogue Scales 26 weeks after implantation | 0, 30, 60, 90, 120, 180, 240
Change in satiety scores as measured by Visual Analogue Scales 52 weeks after implantation | 0, 30, 60, 90, 120, 180, 240
Change in satiety scores as measured by Visual Analogue Scales 3 weeks after explantation | 0, 30, 60, 90, 120, 180, 240
Change in postprandial insulin secretion from baseline 1 week after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial insulin secretion from baseline 26 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial insulin secretion from baseline 52 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial insulin secretion from baseline 3 weeks after explantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucagon secretion 1 week after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucagon secretion 26 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucagon secretion 52 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucagon secretion 3 weeks after explantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucose from baseline 1 week after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucose from baseline 26 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucose from baseline 52 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucose form baseline 3 weeks after explantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial PYY from baseline 1 week after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial PYY from baseline 26 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial PYY from baseline 52 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial PYY from baseline 3 weeks after explantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial ghrelin from baseline 1 week after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial ghrelin from baseline 26 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial ghrelin from baseline 52 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial ghrelin from baseline 3 weeks after explantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucosedependent insulinotropic peptide (GIP) from baseline 1 week after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucosedependent insulinotropic peptide (GIP) from baseline 26 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucosedependent insulinotropic peptide (GIP) from baseline 52 weeks after implantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes
Change in postprandial glucosedependent insulinotropic peptide (GIP) from baseline 3 weeks after explantation | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240 minutes

OTHER OUTCOMES:
Change in gut microbiota as measured by DNA sequencing from baseline | 52 weeks
Change in body composition from baseline 26 weeks after implantation | 1
Change in body composition from baseline 52 weeks after implantation | 1
Change in caloric intake as measured by ad libitum meal test 1 week after implantation | 30 minutes
Change in caloric intake as measured by ad libitum meal test 26 weeks after implantation | 30 minutes
Change in caloric intake as measured by ad libitum meal test 52 weeks after implantation | 30 minutes
Change in caloric intake as measured by ad libitum meal test 3 weeks after explantation | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, Ph.D., Principal Investigator — Center for Diabetes Research, Gentofte Hospital, University of Copenhagen; Ulrich Rohde, MD, Principal Investigator — Center for Diabetes Research, Gentofte Hospital, University of Copenhagen
Locations (1):
- Center for Diabetes Research, Gentofte Hospital, University of Copenhagen, Hellerup, Denmark